CLINICAL TRIAL: NCT06505694
Title: A Clinical Trial to Assess the Impact of an Alcohol Alternative Herbal Tincture on Signs of Stress Anxiety and Sleep Quality.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apothekary (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20381
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Stress
Keywords: Sleep Quality; Sleep Tracker; Relaxation; Herbal Tincture
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double-blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product Arm (Experimental): Participants in this arm will receive the test product, which is an alcohol alternative herbal tincture. The intervention includes taking 2 ml of the test product directly onto the tongue every evening, 1-2 hours before bedtime, for a duration of 8 weeks.
  Interventions: Dietary Supplement: Alcohol Alternative Herbal Tincture (Test Product)
- Placebo Arm (Placebo Comparator): Participants in this arm will receive a placebo. The intervention includes taking 2 ml of the placebo directly onto the tongue every evening, 1-2 hours before bedtime, for a duration of 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alcohol Alternative Herbal Tincture (Test Product) — The test product contains organic vegetable glycerin, distilled water, organic elderberries, organic bilberries, organic beetroot juice powder, organic California poppy (whole plant), organic tart cherry, organic hawthorn berries, organic blue vervain (aerial parts), organic ceylon cinnamon bark, organic black pepper fruit, and L-theanine.
  Arms: Test Product Arm
Dietary Supplement: Placebo — The placebo is designed to match the test product in appearance and taste but does not contain the active herbal ingredients. Participants will take 2 ml of the placebo directly onto the tongue every evening, 1-2 hours before bedtime, for a duration of 8 weeks. The placebo contains organic vegetable glycerin, distilled water, organic beet juice powder, organic tart cherries, organic ceylon cinnamon chips, and natural green food coloring (derived from spirulina and turmeric).
  Arms: Placebo Arm

SUMMARY:
This is a virtual randomized placebo-controlled double-blind trial lasting eight weeks. The trial will assess the effects of a test product on improving sleep quality, promoting a sense of calm, and reducing feelings of stress and anxiety, using a sleep tracker and subject-specific questionnaires. The study involves 80 participants who experience sleep issues and feelings associated with stress and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-65 years
* Male or female
* Good general health
* Experience daily feelings of stress and anxiety within the past two weeks
* Experience daily problems with sleeping, reduced energy levels, and fatigue over the past two weeks
* Have used alcohol products to help relax or sleep within the past two weeks
* Experience tension in the body within the past two weeks
* Experience problems with relaxing in the evening within the past two weeks
* Willing to abstain from alcohol for the duration of the study
* Willing to maintain stable use of other herbal supplements, over-the-counter medications, or prescriptions during the study

Exclusion Criteria:

* Chronic health conditions, including oncological and psychiatric disorders
* Taking SSRIs, sedative, or blood pressure-lowering medications
* Pregnant, breastfeeding, or planning to conceive within the next three months
* Currently enrolled or planning to enroll in another research trial over the next eight weeks
* History of substance abuse
* Known serious allergic reactions requiring an Epi-Pen

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Improvements in Sleep Quality and Mental Well-Being | Baseline, Week 2, Week 4, Week 6, and Week 8
  Changes in sleep quality, mental well-being, stress, and feelings of anxiety will be assessed using self-assessment questionnaires. Participants will complete these questionnaires at specified intervals throughout the study to evaluate the effectiveness of the herbal tincture compared to the placebo.

SECONDARY OUTCOMES:
Changes in Sleep Length and Quality | Baseline, Week 4, and Week 8
  Changes in sleep length and quality will be monitored using a Fitbit sleep tracker. The sleep tracker will collect data on various sleep parameters, including total sleep time and sleep stages, to assess the impact of the herbal tincture compared to the placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No